CLINICAL TRIAL: NCT04782895
Title: A Randomized, Single-blind Study to Compare Immunogenicity of a Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58) Vaccine(E.Coli) (Xiamen Innovax Biotech Co.,Ltd.) Versus Gardasil®9 (Merck & Co., Inc.) in Healthy Females 18-26 Years of Age
Brief Title: Immunogenicity of a Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58)Vaccine(E.Coli) Versus Gardasil®9 in Healthy Females 18-26 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Zhang, professor, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HPV-PRO-011
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cervical Cancer; Condylomata Acuminata
Keywords: human papillomavirus vaccine; immunogenicity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58) Vaccine(E.Coli) group (Experimental): Subjects would receive 3 doses of 270μg/0.5ml Recombinant HPV nonavalent (Types 6/11/16/18/31/33/45/52/58) Vaccine(E.Coli) .
  Interventions: Biological: Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58 )Vaccine(E.Coli)
- Gardasil®9 group (Active Comparator): Subjects would receive 3 doses of 270μg/0.5ml Gardasil®9 .
  Interventions: Biological: Gardasil®9

INTERVENTIONS:
Biological: Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58 )Vaccine(E.Coli) — Three doses administered intramuscularly at 0, 45 day and 6 month.
  Arms: Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58) Vaccine(E.Coli) group
Biological: Gardasil®9 — Three doses administered intramuscularly at 0, 45 day and 6 month.
  Arms: Gardasil®9 group

SUMMARY:
This study is designed to compare the immunogenicity of a novel recombinant human papillomavirus vaccine (types 6,11,16,18,31,33,45,52,58 )(E.Coli) manufactured by Xiamen Innovax Biotech CO., Ltd., with Gardasil®9 in females 18-26 Years of Age.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is female, between and including 18-26 years of age at the first vaccination;
2. Subject is able to understand and comply with the requirements of the protocol(e.g. biological specimen collection, completion of the diary cards, return for follow-up visits), and written informed consent must be obtained from the subject prior to enrollment;
3. Subject who agrees to practice effective contraception within 8 months after the first vaccination or has undergone tubal ligation,subtotal hysterectomy for benign lesion, ovarian benign tumor resection;
4. No previous history of sexually transmitted diseases (including syphilis, gonorrhea, chancroid, venereal lymphogranuloma, groin granuloma, etc.);
5. No previous history of abnormal cervical screening results or cervical intraepithelial neoplasia (CIN);

Exclusion Criteria:

1. Axillary temperature > 37.0℃;
2. Subject who has a positive urine pregnancy test, or is pregnant or breastfeeding;
3. Subject has used of any investigational or non-registered product (drug or vaccine) within 30 days preceding the first dose of study vaccine or plans to use during the study period , or has participated in another clinical research in the past two years, or plans to participate in another research during the study period;
4. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs or systemic corticosteroids (Except intranasal steroid, the use of low dose topical, ophthalmic and inhaled steroid preparations will be permitted.) within 6 months prior to vaccination.
5. Administration of immunoglobulin and/or blood products within 3 months prior to vaccination or planned to use them within 7 months after the first dose.
6. Administration of inactivated vaccine within 14 days prior to vaccination or live vaccine within 21 days;
7. Fever (Axillary temperature ≥38.0℃) 3 days prior to vaccination or system administration of antibiotics or antiviral agents within 5 days prior to vaccination;
8. Subject has received other HPV vaccines or participated in clinical research related to HPV or cervical cancer previously;
9. Subject has immunodeficiency disease, primary disease of important viscera, cancer and autoimmune disease (including systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy due to any condition, and other immunological diseases that investigators believe may influence the immune response).
10. History of severe allergy (e.g., anaphylaxis, generalized urticaria, dyspnea, angioedema, and other significant reaction) to any previous vaccination, or be allergic to any of the components of the study vaccines.
11. Asthma, which has been unstable for the past two years and requires emergency treatment, hospitalization, oral or intravenous corticosteroids;
12. Subject has Serious medical disorders;
13. Self-report coagulation disorders or abnormal coagulation function;
14. Epilepsy, excluding febrile epilepsy under 2 years of age, alcoholic epilepsy 3 years prior to abstinence or simple epilepsy that does not require treatment in the past 3 years;
15. Medical, psychological, social conditions, occupation or other factors, which considered by the investigator that may influence the conduct of the clinical study.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 488 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 type specific neutralizing antibody level | 7 months after the first dose
  Anti-HPV 6,11,16,18,31,33,45,52 and 58 seroconversion rates and geometric mean concentrations at months 7

SECONDARY OUTCOMES:
safety1:Local and systematic adverse events/reactions occurred within 7 days after each vaccination. | During the 7-day period following each vaccination
  Local and systematic adverse events/reactions occurred within 7 days after each vaccination.
safety2:Adverse events/reactions occurred within 30 days after each vaccination. | Within 30 days (Day 0-30) after any vaccination
  Adverse events/reactions occurred within 30 days after each vaccination.
safety3:Severe adverse events occurred throughout the study. To evaluate number of SAEs compared with the control vaccine. | Up to 8 month
  Severe adverse events occurred throughout the study. To evaluate number of SAEs compared with the control vaccine.
safety4:Pregnancy and pregnancy outcome. To evaluate number of births and terminations compared with the control vaccine. | Up to 8 month
  Pregnancy and pregnancy outcome. To evaluate number of births and terminations compared with the control vaccine.

OTHER OUTCOMES:
Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 type specific IgG antibody level | 7 months after the first dose
  Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 seroconversion rates and geometric mean concentrations at months 7(type specific IgG antibody)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, master, Study Chair — Xiamen University; Feng-cai Zhu, master, Principal Investigator — Jiangsu Provincial Centre for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Centre for Disease Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhu FC, Zhong GH, Huang WJ, Chu K, Zhang L, Bi ZF, Zhu KX, Chen Q, Zheng TQ, Zhang ML, Liu S, Xu JB, Pan HX, Sun G, Zheng FZ, Zhang QF, Yi XM, Zhuang SJ, Huang SJ, Pan HR, Su YY, Wu T, Zhang J, Xia NS. Head-to-head immunogenicity comparison of an Escherichia coli-produced 9-valent human papillomavirus vaccine and Gardasil 9 in women aged 18-26 years in China: a randomised blinded clinical trial. Lancet Infect Dis. 2023 Nov;23(11):1313-1322. doi: 10.1016/S1473-3099(23)00275-X. Epub 2023 Jul 17. PMID 37475116